CLINICAL TRIAL: NCT04440124
Title: Does the Incremental Shuttle Walk Test Predict the Development of a Hospital Acquired Pneumonia in Patients Undergoing Elective Oesophagectomy: A Prospective Cohort Study
Status: Completed | Type: Observational
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, David McWilliams, Consultant Physiotherapist, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: JW01
Record Dates: First submitted 2020-06-14; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Oesophageal Cancer
Keywords: physiotherapy; shuttle walk test; hospital acquired pneumonia; outcomes; oesophagectomy
MeSH Terms: conditions — Esophageal Neoplasms; Healthcare-Associated Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Incremental shuttle walk test — All patients were reviewed by a physiotherapist during their pre-assessment clinic one week prior to surgery to complete an incremental shuttle walk test (ISWT). The ISWT was completed according to a standardised protocol and involved patients walking around 2 cones set up 9 metres apart. Patients were asked to cover the distance between the cones in time to auditory cues. Oxygen levels and heart rate were recorded during the assessment with the use of a portable pulse oximeter. The test was stopped when patients could no longer keep pace with the auditory cues or were too breathless to continue. The total distance mobilised was recorded.

SUMMARY:
The purpose of this study was to assess the predictive value of the incremental shuttle walk test on rates of hospital acquired pneumonia for patients undergoing oesophagectomy.

DETAILED DESCRIPTION:
Field tests to objectively measure functional capacity are becoming of greater importance when looking to assess an individual's fitness for surgery. One such field test is the incremental shuttle walk test (ISWT). An externally paced, maximal excursion test, the ISWT is a simple and easily reproducible test that is widely used within cardiac and pulmonary populations and shown to correlate well with Vo2 mas on a cardiopulmonary exercise test. Previous studies looking at the benefit of the ISWT in predicting post-operative outcomes within the oesophagastric population have demonstrated that walking less than 350 meters has been associated with significantly higher rates of mortality at 30 days and 3 years. No correlation between ISWT and postoperative respiratory complications in this surgical population has been previously reported.

This study aims to assess whether walking <350 meters on an ISWT predicts the development of hospital acquired pneumonias following an elective oesophagectomy

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with a diagnosis of oesophagogastric cancer listed for an elective oesophagectomy at a large UK tertiary hospital

Exclusion Criteria:

* Patients who were unable to complete the walking test
* patients deemed not fit for surgery
* patients with a significant neurological event peri or post operatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing oesophagectomy
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Hospital acquired pneumonia | during hospital stay, on average 14 days
  The incidence of hospital acquired pneumonia as defined by the US centres for Disease Control

SECONDARY OUTCOMES:
30 day Mortality | 30 days after date of surgery
  Mortality rates 30 days post operatively
90 day Mortality | 90 days following date of surgery
  Mortality rates 90 days post operatively

CONTACTS AND LOCATIONS:
Locations (1):
- UHB NHS Foundation Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No